CLINICAL TRIAL: NCT07152314
Title: Digital Quantification of Dental Plaque Based on Intraoral Scanner Images
Status: Not yet recruiting | Type: Observational
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, MOHAMED AHMED HASSAN, Professor, University of Guarulhos
Other Study IDs: 85446624.8.0000.5506
Record Dates: First submitted 2025-08-21; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Dental Plaque (Diagnosis); Dental Plaque Imaging Methods; Dental Plaque; Gingivitis; Periodontal Disease
Keywords: Dental Biofilm; Intraoral Scanner; Preventive Dentistry; Plaque quantification; Digital Diagnosis
MeSH Terms: conditions — Dental Plaque; Disease; Gingivitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Digital plaque quantification using intraoral scanner — Participants will undergo three-dimensional intraoral scanning at three time points during a single session: initial scanning (T0), after biofilm disclosure with plaque disclosing solution (T1), and after supervised toothbrushing (T2).

SUMMARY:
This diagnostic validation study aims to develop and validate a digital method for dental biofilm quantification using three-dimensional images obtained by an intraoral scanner. Twenty participants will undergo intraoral scanning at three time points: before and after plaque disclosure, and after supervised toothbrushing. The digital method's accuracy will be compared with traditional clinical assessment methods (Turesky Plaque Index).

DETAILED DESCRIPTION:
A prospective, evaluator-blinded clinical study including 20 participants (18-65 years) with at least 20 natural teeth and a visible plaque index >20%. Participants will be evaluated at three time points in a single session using TRIOS 4 intraoral scanner. Digital analysis will be performed using Geomagic Control X software to calculate the percentage of surface area covered by plaque. The study includes standardized intraoral photographs and supervised toothbrushing procedures. This digital method aims to provide a more objective and precise assessment of dental biofilm, overcoming limitations of conventional visual assessment methods.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 20 natural teeth
* Visible plaque index > 20% at initial assessment
* Age between 18 and 65 years
* Both sexes eligible

Exclusion Criteria:

* Use of fixed orthodontic appliances
* Presence of extensive restorations or fixed dentures on the anterior teeth
* Systemic conditions that interfere with the formation of dental biofilm
* Use of medications that alter salivary flow

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will be carried out through different communication channels, including informative posters distributed in the dental clinics of UnG, digital dissemination on the university's official website and its institutional social networks, direct invitation to patients who are on the waiting list of the periodontics clinic, and dissemination by the professors of the undergraduate and graduate clinics. All promotional materials will clearly state the inclusion and exclusion criteria, as well as provide contact information for scheduling, initial screening, and the ethics committee approval number. All participants will attend the Center for Clinical Studies of Univeritas UnG.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Correlation between digital 3D intraoral scans and traditional plaque assessment methods | Single session (approximately 1.5-2 hours)
  Correlation between the percentage of dental surface area covered by biofilm quantified by the digital method (intraoral scanner) and the plaque index obtained by the traditional clinical method (Quigley-Hein Plaque Index modified by Turesky)

SECONDARY OUTCOMES:
Correlation between digital 2D images and traditional plaque assessment methods | Single session (approximately 1.5-2 hours)
  Correlation between the percentage of dental surface area covered by biofilm quantified by intraoral photographs with different filters and the plaque index obtained by the traditional clinical method (Quigley-Hein Plaque Index modified by Turesky)
Fluorescence imaging capabilities | Single session (approximately 1.5-2 hours)
  Detection sensitivity for plaque, correlation with clinical findings, and reproducibility of fluorescence measurements.
Plaque volume changes analysis | Single session (approximately 1.5-2 hours)
  Ability of the digital method to detect changes in the amount of biofilm, evaluated by the percentage difference in area covered between T0 (initial), T1 (after disclosure) and T2 (after professional brushing).
Plaque thickness changes analysis | Single session (Approximately 1.5-2 hours)
  Ability of the digital method to detect changes in the amount of biofilm, evaluated by the color map difference in area covered between T0 (initial), T1 (after disclosure), and T2 (after professional brushing), and correlating those with other features, such as disclosing agent color and fluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hassan, PhD, Principal Investigator — University of Guarulhos
Locations (1):
- University of Guarulhos, Guarulhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD will be available for sharing based on a reasonable request

REFERENCES:
- [Background] Del Rey YC, Rikvold PD, Johnsen KK, Schlafer S. A fast and reliable method for semi-automated planimetric quantification of dental plaque in clinical trials. J Clin Periodontol. 2023 Mar;50(3):331-338. doi: 10.1111/jcpe.13745. Epub 2022 Nov 28. PMID 36345833

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT07152314/Prot_SAP_ICF_000.pdf